CLINICAL TRIAL: NCT00657735
Title: A Prospective Double Blind Randomized Controlled Trial To Explore The Tolerability, Safety And Efficacy Of The H1-Coil Deep Transcranial Magnetic Stimulation (TMS) In Subjects With Bipolar Depression
Brief Title: Double Blind Randomized Controlled, H1 Coil In Subjects With Bipolar Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shalvata Mental Health Center (Other)
Collaborators: Brainsway (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BR-BIP-02
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Bipolar Depression
Keywords: bipolar; depression; prefrontal; cortex; antidepressant; response
MeSH Terms: conditions — Bipolar Disorder; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Deep TMS treatment
  Interventions: Device: H-Coil deep TMS
- 2 (Sham Comparator): inactive stimulation
  Interventions: Device: sham

INTERVENTIONS:
Device: H-Coil deep TMS — 20 daily deep rTMS treatments
  Other Names: H1 coil dTMS
  Arms: 1
Device: sham — inactive treatment
  Arms: 2

SUMMARY:
The purpose of the study is to explore the efficacy and safety of H1-Coil deep brain rTMS in subjects with bipolar depression , currently treated with mood stabilizer and previously unsuccessfully treated with antidepressant medications

ELIGIBILITY:
Inclusion Criteria:• Outpatients

* Diagnosed by two senior psychiatrists as suffering from bipolar depression (BP1, BP2) episode according to DSM IV using the Structured Clinical Interview for DSM-4 (SCID), with additional requirement of duration for the current episode ≥ 4 weeks and CGI ≥ 4.
* Rating on HAM-D (17 items) >20 and item 1 ≥2 at the screening visit.
* Age: 18-65 years.
* Gave informed consent for participation in the study.
* Negative answers on safety screening questionnaire for transcranial magnetic stimulation
* Taking mood stabilizing medication (e.g., lithium) on an acceptable range of dosage according to recent blood examination or antipsychotic medication as mood stabilizers prescribed by their treating physician
* According to the treating physician the patient is compliant in taking the mood-stabilizing medication.
* Medication resistance to at least two different antidepressant treatments, defined as resistance to a minimum of 2 antidepressant drug trials of adequate dose and duration in the current episode or previous episodes defined as a minimum level of 3 on the ATHF per antidepressant drug-trial.
* Patients who have not completed antidepressant trials of adequate dose and duration due to intolerance to therapy may be included if they have demonstrated intolerance to 3 or more anti-depressant medications in the current or a previous episodes.
* If currently taking antidepressant pharmacotherapy, must be clinically appropriate to discontinue treatment with those agents.
* Able to tolerate psychotropic medication washout and no psychotropics during the H-coil deep brain rTMS other than benzodiazepine at equivalent dose of up to 3 mg lorazepam every day.
* Right hand dominance.

Exclusion Criteria:• Diagnosis as suffering from other diagnosis on axis 1 (like: schizophrenia, geriatric depression).

* Diagnosis as suffering from Severe Borderline Personality Disorder or hospitalized due to exacerbation related to of borderline personality disorder.
* Substantial suicidal risk as judged by the treating psychiatrist.
* Attempted suicide in the past year.
* Patients with a bipolar cycle of less than 30 days.
* History of epilepsy or seizure in first degree relatives.
* History of head injury.
* History of any metal in the head (outside the mouth).
* Known history of any metallic particles in the eye, implanted cardiac pacemaker or any intracardiac lines, implanted neurostimulators, surgical clips or any medical pumps.
* History of frequent or severe headaches.
* History of migraine.
* History of hearing loss.
* Known history of cochlear implants
* History of substance abuse within the past 6 months (except nicotine and caffeine) or alcoholism
* Pregnancy or not using a reliable method of birth control.
* Unstable Systemic and metabolic disorders.
* Unstable neurological or medical disease
* Inadequate communication with the patient.
* Under custodial care.
* Participation in current clinical study or clinical study within 30 days prior to this study.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
change in the Hamilton depression rating scale score | 7 weeks

SECONDARY OUTCOMES:
Clinical antidepressant remission at the end of the treatment, defined as exit Hamilton Depression Rating Scale <10. | 7 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- shalvataMHC, Hod HaSharon, Israel